CLINICAL TRIAL: NCT05079737
Title: A Sample Collection Study to Assess the Prevalence of Gene Mutations Associated With Photoaging in Facial Skin From Adults: Establishing Population Norms
Brief Title: Sample Collection Study to Assess Prevalence of Gene Mutations: Establishing Population Norms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DermTech (Other)
Responsible Party: Sponsor
Other Study IDs: DermTech 21-02
Record Dates: First submitted 2021-09-09; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Photoaging

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Skin samples collected non-invasively from the face using the DermTech non-invasive sample collection kit will be collected and stored for future DNA mutation assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with Fitzpatrick Skin Type I-III: Subjects 21 years of age or older with Fitzpatrick Skin Type I-III will be enrolled and analyzed by age.
  Interventions: Other: Mutation Burden
- Subjects with Fitzpatrick Skin Type IV-VII: Subjects 21 years of age or older with Fitzpatrick Skin Type IV-VII will be enrolled and analyzed by age.
  Interventions: Other: Mutation Burden

INTERVENTIONS:
Other: Mutation Burden — Subjects will have their facial samples analyzed for DNA mutation burden.

SUMMARY:
This is a multi-center, sample collection study to quantitatively assess the presence of gene mutations in subject's skin collected non-invasively. Subjects who consult with a dermatologist or other clinicians will be approached for participation in the study. Once IRB approved informed consent is obtain, subject demographic information, history of sun exposure and samples will be collected.

DETAILED DESCRIPTION:
This is a multi-center, sample collection study to quantitatively assess the presence of gene mutations in subject's skin collected non-invasively. Subjects who consult with a dermatologist or other clinicians will be approached for participation in the study. Once confirmation of participation is confirmed subjects will undergo the informed consent process.

Once consented the subject will have their medical history reviewed, concomitant medications and demographic information recorded, complete a sun-exposure questionnaire, have photoaging characteristics (such as melasma, wrinkles, AK lesion(s)) recorded, record their assessment of photoaging, have skin samples collected non-invasively and complete the local skin reaction and local tolerability assessments. A select number of subjects will also have a facial photograph taken.

If the location to be sampled contains a lesion, then the collection should occur as close as possible to the target area. The site staff and/or subject will be responsible for collecting the skin samples.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 21 years of age presenting to the clinic for medical consultation;
2. In good health, determined by no clinically significant findings from medical history,
3. Willing to complete all study procedures required by the protocol; and
4. Willing to provide informed consent to participate in this trial.

Exclusion Criteria:

1. Have any skin disorder including acne, rosacea, psoriasis, atopic dermatitis and active skin cancer(s) that appear in the facial area where sample collection will be taken and could confound the results of the trial;
2. Has a suspicious lesion (i.e., actinic keratosis lesion) in an area that is expected to be sampled and requires further medical follow-up,
3. Pregnant or breast feeding,
4. Hospitalization within 4 weeks before enrollment,
5. Previously provided samples for this study,
6. Receipt of any investigational drug therapy within four weeks of study enrollment, or concurrent participation in another interventional clinical study,
7. Documented substance abuse, any other significant medical condition that would indicate an unreasonable risk to the potential study participate or potential interference with the procedures, or would negatively affect the study subject's reliability and compliance with the study schedule of events, and
8. Chemical peel or treatment with a laser in the facial area within 3 months prior to enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to approximately 5,000 adults presenting to clinics for consultations will be enrolled into this study.
  Subjects will be enrolled across a wide range of demographics and age ranges. A minimum of 3000 subjects of Fitzpatrick Skin Type I-III skin types (Group 1) and 1000 subjects of Fitzpatrick IV-VI (Group 2) will be enrolled. This will include, but is not limited to races such as Caucasian, African American, and subjects of Asian descent. At least 100 subjects per Fitzpatrick Skin Type group will be from the following age ranges; 21-30, 31-40, 41-50, 51-60 and >61 will be enrolled.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence rate of mutations | 1 day
  The prevalence rate of selected DNA mutations will be quantitated

SECONDARY OUTCOMES:
Correlate gene mutations with demographic information | 1 day
  prevalence of mutations relative to age, sex, race and ethnicity
Correlation gene mutation with sun exposure scores | 1 day
  prevalence of mutations relative to life time sun exposure

CONTACTS AND LOCATIONS:
Overall Officials: Loren Clarke, MD, Study Director — DermTech
Locations (1):
- West Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided